CLINICAL TRIAL: NCT06574269
Title: A Phase 2, Open-label, Dose-escalation Study to Evaluate Pharmacokinetics, Pharmacodynamics, Bioavailability, Safety, and Tolerability of TLC590 in Multiple Surgical Models
Brief Title: A Study on TLC590 for Managing Postsurgical Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TLC Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Taiwan Liposome Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLC590A2006
Record Dates: First submitted 2024-08-25; First posted 2024-08-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Postsurgical Pain Management
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1, Cohort 1 (Experimental): Bunionectomy: Increasing dose cohorts for TLC590
  Interventions: Drug: TLC590
- Part 1, Cohort 2 (Experimental): Laparoscopy-assisted Open Ventral Hernia: TLC590
  Interventions: Drug: TLC590
- Part 2, Cohort 3 (Experimental): Breast Augmentation: TLC590 or Ropivacaine
  Interventions: Drug: TLC590; Drug: Ropivacaine
- Part 2, Cohort 4 (Experimental): Breast Augmentation: TLC590 or Ropivacaine
  Interventions: Drug: TLC590; Drug: Ropivacaine
- Part 2, Cohort 5 (Experimental): Breast Augmentation: TLC590 with the SMC-suggested dose
  Interventions: Drug: TLC590
- Part 3, Cohort 6 (Experimental): Laparoscopy-assisted Open Ventral Hernia: The MTD of TLC590
  Interventions: Drug: TLC590
- Part 3, Cohort 7 (Experimental): Total Knee Arthroplasty: The MTD of TLC590
  Interventions: Drug: TLC590
- Part 3, Cohort 8 (Experimental): Abdominoplasty: The MTD of TLC590
  Interventions: Drug: TLC590

INTERVENTIONS:
Drug: TLC590 — Sequentially enrolled into increasing dose cohorts from low to high to receive a dose of TLC590
  Other Names: TLC590 (Ropivacaine Extended-Release Injectable Suspension)
  Arms: Part 1, Cohort 1
Drug: TLC590 — TLC590 Dose 1
  Other Names: TLC590 (Ropivacaine Extended-Release Injectable Suspension)
  Arms: Part 2, Cohort 3
Drug: TLC590 — TLC590 Dose 2
  Other Names: TLC590 (Ropivacaine Extended-Release Injectable Suspension)
  Arms: Part 2, Cohort 4
Drug: TLC590 — The MTD of TLC590
  Other Names: TLC590 (Ropivacaine Extended-Release Injectable Suspension)
  Arms: Part 3, Cohort 6; Part 3, Cohort 7; Part 3, Cohort 8
Drug: TLC590 — TLC590 Dose 3 (The SMC-suggested dose)
  Other Names: TLC590 (Ropivacaine Extended-Release Injectable Suspension)
  Arms: Part 2, Cohort 5
Drug: Ropivacaine — Ropivacaine
  Other Names: Ropivacaine HCL Injection
  Arms: Part 2, Cohort 3; Part 2, Cohort 4
Drug: TLC590 — TLC590
  Other Names: TLC590 (Ropivacaine Extended-Release Injectable Suspension)
  Arms: Part 1, Cohort 2

SUMMARY:
This Phase 2 open-label trial investigates the pharmacokinetics (PK), pharmacodynamics, and safety profile of TLC590 across various surgical procedures. Researchers aim to determine the maximum tolerated dose (MTD) of TLC590 via Safety Monitoring Committee (SMC).

The study evaluates TLC590 in bunionectomy, laparoscopy-assisted open ventral hernia repair, breast augmentation, abdominoplasty, and total knee arthroplasty models. Additionally, it determines the relative bioavailability of TLC590 to ropivacaine injection.

DETAILED DESCRIPTION:
This Phase 2, open-label, multi-center study is a 3-part study to be performed in approximately 120 subjects undergoing multiple surgical procedures receiving TLC590 or ropivacaine injection. Subjects eligible based on inclusion and exclusion criteria will receive study drug administered via infiltration. Subjects entering all parts of the study will undergo the consent and screening procedures, eligibility requirements, and PK and safety evaluations during their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent
2. Male or female aged 18 to 70 years, inclusive. For the Part 2 breast augmentation surgical model, only females can be enrolled
3. Scheduled to undergo one of the following elective surgeries, with no additional procedures and be able to use the anesthesia regimen:

   1. Unilateral first metatarsal bunionectomy (Cohort 1)
   2. Laparoscopy-assisted open ventral hernia repair (Cohort 2 and 6)
   3. Breast augmentation (Cohort 3 through 5)
   4. Unilateral total knee arthroplasty (Cohort 7)
   5. Abdominoplasty (tummy tuck) (Cohort 8)
4. ASA Physical Status Classification of 1 or 2
5. Male subjects must be either biologically or surgically sterile or commit to the use of a reliable method of birth control (must agree to use double-barrier contraception in the event of sexual activity) or be practicing abstinence for the duration of the study and for 30 days after study drug administration
6. Female subjects are eligible only if all the following apply:

   1. Not pregnant with a negative serum pregnancy test at Screening and negative urine pregnancy test on Day 1 before surgery (pregnancy test not required for females of non-childbearing potential, defined as surgically sterile or post-menopausal)
   2. Not lactating
   3. Not planning to become pregnant during the study
   4. If of childbearing potential, commits to the use of a highly effective method of birth control for the duration of the study and or at least 30 days after study drug administration
7. BMI >18 ~ ≤39 kg/m2

Exclusion Criteria:

1. A clinically significant abnormal clinical laboratory test value
2. Evidence of a clinically significant 12-lead ECG
3. History of orthostatic hypotension, syncope, or other syncopal attacks
4. History or any clinical manifestation of significant renal, hepatic, gastrointestinal, cardiovascular, metabolic, neurologic, psychiatric, or other condition that has been assessed by the Investigator to be unsuitable for participation in the study
5. History of seizures or taking anticonvulsants during the Screening period
6. History of cardiac arrhythmia or taking Class III antiarrhythmic drugs including amiodarone, dofetilide, dronedarone, sotalol, or ibutilide during the Screening period
7. History of sleep apnea or on home CPAP treatment
8. History of hypersensitivity to ropivacaine, any other amide-type local anesthetic, propofol, hydromorphone, fentanyl, midazolam, acetaminophen, oxycodone, or morphine (or other opioids)
9. History of severe or refractory PONV due to other etiologies, including, but not limited to gastric outlet obstruction, hypercalcemia, or active peptic ulcer, deemed clinically significant by the Investigator
10. Any lifetime history of a suicidal attempt or any suicidal behavior, as assessed by the C-SSRS at Screening
11. History or positive test results of HIV, HCV, or HBV
12. History or current report of substance abuse including illicit drug abuse and/or alcohol abuse (regularly drinks >4 units of alcohol per day: 1 unit = 8 oz. beer, 3 oz. wine, or 1 oz. spirits) within 2 years prior to Screening
13. Positive results on the urine drug screen or alcohol breath test indicative of illicit drug or non-prescribed drug or alcohol abuse at Screening or on Day 1 before surgery. Prescribed medication that is known to result in a positive drug test is allowed. Marijuana (medical or recreational) is not allowed
14. Pre-existing concurrent acute, or chronic painful restrictive/physical condition that may confound postoperative pain assessments or is expected to require analgesic treatment during the study
15. Has known or suspected daily use of opioids for longer than 4 days per week within the previous 6 months prior to Screening
16. Is taking daily analgesics for longer than 4 days per week for a chronically painful condition during the Screening period. Not exclusionary if it is utilized for pain related to the total knee arthroplasty indication
17. Is receiving oxygen therapy during the Screening period
18. Use of any of the following medications within 5 half-lives prior to the study surgical procedure or as specified
19. Malignancy in the last 2 years prior to Screening, except for non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix
20. Personal or family history of malignant hyperthermia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To determine the relative bioavailability of TLC590 compared to ropivacaine HCl injection (Part 2) | 0-168 hours
To determine the MTD of TLC590 in subjects with breast augmentation surgery (Part 2) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Tien-Tzu Tai, MD, Study Director — Taiwan Liposome Company
Locations (2):
- United States (2):
  - First Surgical Hospital, Bellaire, Texas
  - Memorial Hermann Village, Houston, Texas